CLINICAL TRIAL: NCT07197567
Title: Evaluation of Equivalent Minimum Alveolar Concentration During General Anesthesia: An Observational Study
Brief Title: Equivalent MAC in General Anesthesia
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Other Study IDs: SEAH-EMAC-2025
Record Dates: First submitted 2025-08-31; First posted 2025-09-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: General Anesthesia; Intraoperative Monitoring; Anesthetic Depth
Keywords: Equivalent Minimum Alveolar Concentration; eMAC; Minimum Alveolar Concentration; MAC; Bispectral Index; BIS; Anesthesia Depth; Combined Intravenous and Inhalational Anesthesia; CIVIA; Propofol; Sevoflurane
MeSH Terms: interventions — Sevoflurane; Remifentanil; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhalational Anesthesia Group: Patients receiving general anesthesia maintained with inhalational agents (e.g., sevoflurane) according to standard clinical practice.
  Interventions: Drug: Sevoflurane + Remifentanil
- Combined Intravenous-Inhalational Anesthesia (CIVIA) Group: Patients receiving general anesthesia with a combination of intravenous and inhalational agents according to standard clinical practice.
  Interventions: Drug: Sevoflurane + Propofol + Remifentanil

INTERVENTIONS:
Drug: Sevoflurane + Remifentanil — Combination of an inhalational anesthetic (sevoflurane) and an intravenous opioid analgesic (remifentanil), both routinely used in clinical practice for maintenance of general anesthesia. These agents are administered according to standard of care, not as experimental interventions.
  Groups: Inhalational Anesthesia Group
Drug: Sevoflurane + Propofol + Remifentanil — Combination of an inhalational anesthetic (sevoflurane), an intravenous anesthetic (propofol), and an intravenous opioid analgesic (remifentanil). These agents are routinely used together in clinical practice for combined intravenous-inhalational anesthesia (CIVIA). All drugs are administered according to standard of care, not as experimental interventions.
  Groups: Combined Intravenous-Inhalational Anesthesia (CIVIA) Group

SUMMARY:
This observational study aims to evaluate the clinical applicability of the Equivalent Minimum Alveolar Concentration (eMAC) parameter during general anesthesia. eMAC is a recently developed index that combines the effects of both inhalational and intravenous anesthetics, providing a unified measure of anesthetic depth. While the traditional Minimum Alveolar Concentration (MAC) is widely used for inhalational agents, it does not reflect intravenous anesthetics or combined techniques such as Combined Intravenous and Inhalational Anesthesia (CIVIA).

In this study, adult patients undergoing elective surgery under general anesthesia will be observed. Standard clinical practice will not be altered. Demographic and clinical parameters, including eMAC, MAC, Bispectral Index (BIS), and hemodynamic variables, will be recorded at defined perioperative time points. No experimental drugs or additional procedures will be administered.

The primary aim is to investigate the correlation between eMAC and MAC values obtained during anesthesia. Secondary objectives include assessing the relationship between eMAC and BIS values, comparing eMAC, MAC, and BIS across different anesthetic techniques, and evaluating hemodynamic stability in relation to anesthetic depth.

The results of this study may contribute to a better understanding of eMAC and its potential role in clinical anesthesia practice.

DETAILED DESCRIPTION:
This is a prospective, observational study designed to evaluate the Equivalent Minimum Alveolar Concentration (eMAC) parameter during general anesthesia. eMAC is a composite index that incorporates the anesthetic effects of both inhalational agents and intravenous anesthetics, such as propofol and remifentanil, allowing assessment of anesthetic depth under combined techniques (CIVIA). While the traditional Minimum Alveolar Concentration (MAC) is well established for inhalational agents, its applicability is limited in cases where intravenous agents are administered. eMAC has been proposed as a more comprehensive measure, but clinical validation is lacking.

Adult patients (ages 18-65, ASA I-III) scheduled for elective surgical procedures under general anesthesia will be enrolled. No experimental interventions will be performed; anesthetic management will follow routine clinical practice. Participants will be observed in three groups, based on the anesthetic technique selected by the attending anesthesiologist.

Data collection will include demographic and baseline clinical variables, as well as anesthetic depth parameters (eMAC, MAC, Bispectral Index [BIS]) and hemodynamic variables (heart rate, mean arterial pressure, SpO₂). Measurements will be recorded at predefined time points: prior to induction (T0), 5 minutes after induction (T1), at the beginning of surgery (T2), at the midpoint of surgery (T3), and at the end of surgery (T4).

The primary outcome measure is the correlation between eMAC and MAC values obtained during anesthesia. Secondary outcome measures include the correlation between eMAC and BIS values, comparisons of eMAC, MAC, and BIS among different anesthetic techniques, and evaluation of hemodynamic stability in relation to anesthetic depth.

Statistical analysis will be performed using appropriate parametric or non-parametric tests, depending on the distribution of variables. Correlation analyses will be conducted using Pearson or Spearman methods, and the impact of demographic factors on eMAC will be explored using multivariate regression. A p-value <0.05 will be considered statistically significant.

The anticipated enrollment is 60 patients. The study is planned to start in September 2025 and is expected to be completed by November 2025. Findings may provide novel insights into the clinical validity of eMAC as a tool for assessing anesthetic depth, and its relationship with established parameters such as MAC and BIS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Scheduled for elective surgery under general anesthesia
* American Society of Anesthesiologists (ASA) Physical Status I-III
* Feasibility of Bispectral Index (BIS) monitoring
* Provision of written informed consent

Exclusion Criteria:

* History of neurological disease (e.g., epilepsy, dementia, severe brain injury)
* Known allergy to anesthetic agents
* Severe cardiovascular or respiratory failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective surgical procedures under general anesthesia at Sakarya University Training and Research Hospital, Department of Anesthesiology and Reanimation, will be considered for enrollment. Patients represent a typical surgical population with ASA physical status I-III.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Correlation between Equivalent Minimum Alveolar Concentration (eMAC) and Minimum Alveolar Concentration (MAC) | From induction of anesthesia until the end of surgery (measured at five perioperative time points: prior to induction, 5 minutes after induction, at surgical incision, at the midpoint of surgery, and at the end of surgery)
  To determine the relationship between eMAC values and conventional MAC values obtained from the anesthesia workstation.

SECONDARY OUTCOMES:
Correlation between eMAC and Bispectral Index (BIS) | From induction of anesthesia until the end of surgery (measured at five perioperative time points: prior to induction, 5 minutes after induction, at surgical incision, at the midpoint of surgery, and at the end of surgery)
  To assess the relationship between eMAC values and BIS as indicators of anesthetic depth.
Comparison of eMAC, MAC, and Bispectral Index (BIS) Values Measured by Anesthesia Workstation and BIS Monitor Across Different Anesthetic Techniques | From induction of anesthesia until the end of surgery (measured at five perioperative time points: prior to induction, 5 minutes after induction, at surgical incision, at the midpoint of surgery, and at the end of surgery)
  To compare anesthetic depth parameters obtained from the anesthesia workstation (eMAC and MAC values) and BIS monitor (BIS values) among patients managed with inhalational anesthesia, total intravenous anesthesia (TIVA), or combined intravenous-inhalational anesthesia (CIVIA).
Heart Rate During Anesthesia | From induction of anesthesia until the end of surgery (measured at five perioperative time points: prior to induction, 5 minutes after induction, at surgical incision, at the midpoint of surgery, and at the end of surgery)
  To evaluate heart rate (beats per minute) in relation to anesthetic depth parameters across study groups.
Mean Arterial Pressure During Anesthesia | From induction of anesthesia until the end of surgery (measured at five perioperative time points: prior to induction, 5 minutes after induction, at surgical incision, at the midpoint of surgery, and at the end of surgery)
  To evaluate mean arterial pressure (mmHg) in relation to anesthetic depth parameters across study groups.
Peripheral Oxygen Saturation (SpO₂) During Anesthesia | From induction of anesthesia until the end of surgery (measured at five perioperative time points: prior to induction, 5 minutes after induction, at surgical incision, at the midpoint of surgery, and at the end of surgery)
  To evaluate peripheral oxygen saturation (percentage, %) in relation to anesthetic depth parameters across study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Tas Tuna, Professor, M.D., Principal Investigator — Sakarya University Faculty of Medicine
Locations (1):
- Sakarya University Training and Research Hospital, Department of Anesthesiology and Reanimation, Sakarya, Adapazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center observational study with a limited sample size, and data contain potentially identifiable clinical information. Only aggregated results will be reported in publications.

REFERENCES:
- [Background] Zhang H, Zhang J, Li X, He S, Deng Z, Wang L, Wang Y, Wang X, Wan C, Huang F, Zhu Z, Dong H. Feasibility Study of an Indicator of Equivalent Potency of Multiple Anesthetics Normalized by Minimum Alveolar Concentration Derived From Response Surface Models. Anesth Analg. 2025 Apr 17. doi: 10.1213/ANE.0000000000007514. Online ahead of print. PMID 40244902